CLINICAL TRIAL: NCT03390699
Title: The Microbial Profile Among Patients Before and After Partial Maxillectomy
Brief Title: Microbial Profile Among Patients Before and After Partial Maxillectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0259-17-RMB CTIL
Record Dates: First submitted 2017-12-28; First posted 2018-01-04 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-12

CONDITIONS: Microbiology, Maxilla

STUDY DESIGN:
Intervention Model Description: Microbial profile among patients before partial maxillectomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- before and after partial maxillectomy (Experimental): Microbial profile among patients before and after partial maxillectomy
  Interventions: Diagnostic Test: Microbial profile

INTERVENTIONS:
Diagnostic Test: Microbial profile — microbiological testing

SUMMARY:
Patients after maxillecotmy develop gum disease and teeth decay often. these two diseases are caused by bacteria. In addition, these patients may have oral infections such as candida . The therapeutic approach now days to these diseases (dental decay and periodontal disease) can change following the results of the study.

the purpose of the study is to examine whether the connection between the oral cavity and anatomical structures exposed by maxillectomy procedure causes a change in the level of microbes examined. To the best of our knowledge, there are not yet studies examined the clinical and microbiological changes in the oral cavity before and after surgery.

DETAILED DESCRIPTION:
This study will include 15 patients who are scheduled to undergo partial maxillectomy as part of a prescribed treatment program prior to their eligibility for the study. The patients will undergo the surgery at the Department of Otolaryngology or Oral and Maxillofacial Surgery and will be given an obturator during surgery by a physician from the Internal and Maxillofacial Rehabilitation Department of the School of Dentistry .

demographic data on the patient's age and gender, general medical history, smoking habits, oral and periodontal and clinical examination (presence of periodontal disease) and microbiological testing will be preformed.

ELIGIBILITY:
Inclusion Criteria:

1. signed Consent form
2. Patients who are supposed to undergo Maxilla removal without closing the defect using a tissue implant and will need to complete the missing area by an obturator.
3. Men and women aged 18 and over

Exclusion Criteria:

1. Allergy to substances from which the obturator is made.
2. Pregnant women
3. Taking antibiotic drugs that affect bacterial flora 4 weeks before taking the saliva sample.
4. Psychiatric problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
microbial types | 6 months
  types of microbes on the sliva

CONTACTS AND LOCATIONS:
Overall Officials: Zvi Gutmacher, DMD, Principal Investigator — Rambam Health Care Campus

IPD SHARING:
Plan to Share IPD: No